CLINICAL TRIAL: NCT04145206
Title: Ankle Instability in Flamenco Dancers
Status: Completed | Type: Observational
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Aurora Castro Mendez, Proffesor, PhD, University of Seville
Other Study IDs: 170111
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Ankle Disease; Dance
Keywords: ankle; dance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: the experimental group is characterized by the practice of flamenco dance
  Interventions: Behavioral: Flamenco dance
- control group: not practice of flamenco dance

INTERVENTIONS:
Behavioral: Flamenco dance — evaluation of ankle injuries in the flamenco dancers
  Groups: experimental group

SUMMARY:
The injuries in the dancers are usually associated with different factors such as the characteristics of the footwear, height of the heel and physical requirements, the articulation of the ankle being the most susceptible when the loads are not adequately dealt. The main objective is to evaluate in a sample of subjects if there is a difference in the stability of the ankle, as a consequence of previous sprains, between flamenco dancers and dancers and a dance-free control group.

DETAILED DESCRIPTION:
An observational study. This study has involved a population of 26 subjects divided into two groups of 13 each is studied (40,15 ± 4,675 años); the experimental group is characterized by the practice of flamenco dance

ELIGIBILITY:
Inclusion Criteria:

Flamenco dancers

-

Exclusion Criteria:

* no

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study has involved a population of 26 healthy subjects divided into two groups of 13 each one
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Ankle drawer test | A day, the inclusion day in the study
  Evaluation of the ankle drawer test, in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Aurora Castro Mendez, Seville, Spain

IPD SHARING:
Plan to Share IPD: No